CLINICAL TRIAL: NCT02797080
Title: Long-Term Safety Extension Study of ACTIMMUNE® (Interferon γ-1b) in Children and Young Adults With Friedreich's Ataxia
Acronym: STEADFAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-ACT-303
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Friedreich's Ataxia
Keywords: ACTIMMUNE; interferon y-1b
MeSH Terms: conditions — Friedreich Ataxia | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- interferon γ-1b (Experimental): ACTIMMUNE® will be administered 3 times per week (TIW) by subcutaneous (SC) injection.
  Interventions: Drug: interferon γ-1b

INTERVENTIONS:
Drug: interferon γ-1b — ACTIMMUNE® will be administered three times per week by subcutaneous injection. The initial dose will be individualized for each participant and will be determined by the investigator, provided that the initial dose does not exceed the maximum tolerated dose in HZNP-ACT-302 (NCT02593773). The investigator may subsequently adjust the dose for any participant if deemed clinically appropriate, provided that the dose does not exceed 100 μg/m².
  Other Names: ACTIMMUNE®

SUMMARY:
The purpose of this long term extension study is to evaluate the long-term safety of ACTIMMUNE® (interferon-γ 1b) in participants with Friedreich's Ataxia (FA).

DETAILED DESCRIPTION:
This is a multi-center, open-label, long-term safety extension study of ACTIMMUNE® in the treatment of FA in children and young adults. Participants who complete 26 weeks of treatment and the Week 28 Follow-Up Visit in HZNP-ACT-302 (NCT02593773) will be eligible to enter this long-term safety extension protocol. The Day 1 Visit of this study (HZNP-ACT-303) occurs on the same day as the Week 28 Follow-Up Visit for HZNP-ACT-302 (NCT02593773). Participants will be required to return for clinic visits at least every 6 months. The treatment duration is open-ended, and treatment will continue until ACTIMMUNE® is commercially available for the treatment of FA in the United States or until the Sponsor decides not to continue development for the treatment of FA.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and child assent, if applicable.
* Completed 26 weeks of treatment and the Week 28 Follow-Up visit in Study HZNP-ACT-302 (NCT02593773).
* If female, the subject is not pregnant or lactating or intending to become pregnant during the study, or within 30 days after the last dose of study drug. Female subjects of child-bearing potential must have a negative urine pregnancy test result at Week 26 of Study HZNP-ACT-302 (NCT02593773) and agree to use a reliable method of contraception throughout the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* If in the opinion of the Investigator, patients have a concomitant disease or condition that could interfere with the conduct of the study or potentially put the subject at unacceptable risk, the subject will be excluded from the study.

Ages: 11 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - University of California, Los Angeles Neurology Clinic, Los Angeles, California
  - University of Florida Clinical Research Center, Gainesville, Florida
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon γ-1b: Subcutaneous (SC) ACTIMMUNE® 3 times a week (TIW) at an individualized dose.
Period: Overall Study
Arm/Group | Interferon γ-1b
Started | 38
Completed | 36
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Interferon γ-1b: SC ACTIMMUNE® TIW at an individualized dose
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (3.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: An adverse event (AE) is any untoward medical occurrence, whether or not the event is considered related to the investigational product. A TEAE is any adverse change from the subject's baseline condition, including any laboratory test value abnormality judged as clinically significant by the investigator, that occurs on or after the date of the first dose of study drug administered at home and throughout the duration of the clinical study, whether the adverse event is considered related to the treatment or not. A serious AE (SAE) is an AE that results in death, is life-threatening, results in persistent or significant disability or incapacity, inpatient hospitalization or prolongation of an existing hospitalization, is a congenital anomaly or birth defect, or other medically important event.
Time Frame: Baseline/Day 1 (Week 28 Follow-Up Visit for Study HZNP-ACT-302 ([NCT02593773]) through end of study; mean (SD) duration of treatment was 99.2 (58.48) days.
Population: Safety Population, defined as all participants who received at least 1 dose of study drug after the Baseline Visit for Study HZNP-ACT-303.
Measure: Number; unit: participants
Arm/Group | Interferon γ-1b
Number analyzed (Participants) | 38
participants
  ≥ 1 TEAE | 21
  ≥ 1 Related TEAE | 7
  ≥ 1 SAE | 0
  ≥ 1 Related SAE | 0
  ≥ 1 TEAE Leading to Discontinuation | 0
  ≥ 1 TEAE Leading to Death | 0

ADVERSE EVENTS:
Time Frame: Baseline/Day 1 (Week 28 Follow-Up Visit for Study HZNP-ACT-302 ([NCT02593773]) through end of study; mean (SD) duration of treatment was 99.2 (58.48) days.
Arm/Group | Interferon γ-1b
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 17/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon γ-1b (N=38)
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Headache (Nervous system disorders) | 4
Fatigue (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2

LIMITATIONS AND CAVEATS:
This study was stopped by the Sponsor because the development of ACTIMMUNE® for the treatment of FA was discontinued after Study HZNP-ACT-301 (NCT02415127) failed to meet its primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT02797080/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT02797080/SAP_001.pdf